CLINICAL TRIAL: NCT06247241
Title: A Phase 2a, Open-Label, First-In-Human, Two-Part, Single And Multiple Ascending Dose Study To Evaluate The Safety, Tolerability, And Efficacy Of VMB-100 In Female Subjects With Moderate Stress Urinary Incontinence
Brief Title: A Phase 2a Study To Evaluate VMB-100 In Females With Stress Urinary Incontinence
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study has not enrolled study participants, and will not start enrolling, due to insufficient funding and is withdrawn from .
Sponsor: Versameb AG (Industry)
Collaborators: PPD Development, LP (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VMB-100-U222
Record Dates: First submitted 2024-01-19; First posted 2024-02-07 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-03

CONDITIONS: Stress Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Intervention Model Description: Single and multiple ascending dose
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VMB-100 administration (Experimental): intrasphincteric injection of VMB-100 in the urethra sphincter
  Interventions: Drug: VMB-100

INTERVENTIONS:
Drug: VMB-100 — VMB-100 is administered as intrasphincteric injection in the urethra sphincter

SUMMARY:
The study drug VMB-100 is an mRNA encoding for IGF-1. It is administered by injection into the urethra sphincter, and taken up by the muscle cells. The IGF-1 acts to promote muscle regeneration in the sphincter, which is expected to improve the function of the sphincter and thereby alleviate incontinence (urinary leakage).

DETAILED DESCRIPTION:
Versameb AG (Sponsor) is developing VMB-100 for the treatment of stress urinary incontinence (SUI), and mixed urinary incontinence (MUI) with a predominant stress component, a common and debilitating condition that significantly impacts quality of life, and for which there are currently no approved pharmacological therapies available in the US.

The drug substance of VMB-100 is a mRNA encoding human insulin-like growth factor-1 (IGF-1). VMB-100 is administered as a transurethral injection into the urinary sphincter muscle. The injected mRNA is taken up by the muscle tissue cells and serves as a template for the translation of the protein IGF-1.

Insulin-like growth factor-1 is secreted into the extracellular space, where it acts to promote muscle regeneration of the urinary sphincter via auto- and paracrine activation of downstream pathways in a localized manner.

The current understanding in urology is that reduced maximum urethral closure pressure (MUCP) is the factor most strongly associated with SUI. This implies that improving function of the closure muscles would have therapeutic merit in both SUI as well as MUI with a predominant stress component.

No treatment which restores the physiology (regenerates the urinary sphincter muscle) is currently available. Given IGF-1's role in regenerating/maintaining muscle tissue women with SUI may benefit from a localized increase in IGF-1 levels in the urinary sphincter to regenerate muscle and restore sphincter function, thus alleviating the incontinence.

ELIGIBILITY:
Main inclusion criteria:

* Pre- or peri-menopausal female subject between 18 and 55 years of age
* Body mass index (BMI) of 19 to 35 kg/m2
* Active SUI of moderate severity for at least 6 consecutive months documented in medical history
* Refractory to standard of care measures
* Must not be pregnant, lactating, or actively trying to become pregnant.

Main exclusion criteria:

* Any concurrent condition or any clinically significant abnormality at Screening which in the opinion of the Investigator may affect the interpretation of safety or efficacy data or which otherwise contradicts participation in a clinical study with VMB-100
* Unwilling to undergo transvaginal sonography or cystoscopy
* Urodynamic detrusor overactivity
* History of urinary urge incontinence of neurogenic etiology.
* History of or planning for pelvic radiation.
* History of use of any bulking agent or Botox to treat SUI in the past 12 month.
* History of urethral sling, anterior prolapse repair, and/or other SUI procedures or surgical procedures affecting continence.
* Taking any medications that are known to have an effect on urinary continence or medications that may exacerbate incontinence

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2029-04 (Estimated)

PRIMARY OUTCOMES:
Safety following VMB-100 administration | from baseline/preinjection through study completion (est average 1 year)
  Adverse Events (AEs)
Safety following VMB-100 administration | immediately after the intervention through study completion (est average 1 year)
  Treatment Emergent Adverse Events (TEAEs)
Safety following VMB-100 administration | immediately after the intervention through study completion (est average 1 year)
  Adverse Events of Special Interest (AESIs)
Tolerability of VMB-100 injection, pain | periprocedurally
  measurement of pain by Visual Analogue Scale (0-10, where 0 is no pain and 10 is the worst pain)
Vital signs following VMB-100 administration | from baseline/preinjection through study completion (est average 1 year)
  heart rate, blood pressure, respiratory rate, body temperature
12-lead ECG following VMB-100 administration | from baseline/preinjection through study completion (est average 1 year)
  P-wave, QRS complex, QTc prolongation
Clinical laboratory measurements following VMB-100 administration | from baseline/preinjection through study completion (est average 1 year)
  change in hematology parameters ( proportion of subjects)
Clinical laboratory measurements following VMB-100 administration | from baseline/preinjection through study completion (est average 1 year)
  change in biochemistry parameters (proportion of subjects)
Clinical laboratory measurements following VMB-100 administration | from baseline/preinjection through study completion (est average 1 year)
  change in urinalysis (proportion of subjects)

OTHER OUTCOMES:
Efficacy; effect on incontinence event frequency | from baseline/preinjection through study completion (est average 1 year)
  bladder diary will record number of incontinence events for 7 days prior to each visit
Efficacy; effect on patient assessment of effect | from baseline/preinjection through study completion (est average 1 year)
  patient reported outcomes questionnaire Patient Global Impression of Severity (PGI-S) for stress urinary incontinence
Efficacy; effect on patient assessment of effect | from baseline/preinjection through study completion (est average 1 year)
  patient reported outcomes questionnaire Patient Global Impression of Improvement (PGI-I ) for stress urinary incontinence
Efficacy; effect on patient assessment of effect | from baseline/preinjection through study completion (est average 1 year)
  patient reported outcomes questionnaire; International Consultation on Incontinence Questionnaire (ICIQ)
Efficacy; effect on patient assessment of effect | from baseline/preinjection through study completion (est average 1 year)
  patient reported outcomes questionnaire Kings Health Questionnaire (KHQ)
Pharmacodynamic evaluation; morphologic changes to the urethra sphincter using transvaginal ultrasound | from baseline/preinjection to week 24
  change in sphincter thickness, measured in millimeters